CLINICAL TRIAL: NCT03739424
Title: Egg Consumption, Skeletal Health, and Cognition in Normal Weight and Obese Children: A Randomized Controlled Trial
Brief Title: Skeletal and Cognitive Effects of Nutrition From Eggs
Acronym: SCENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, Dr. Richard D. Lewis, UGA Foundation Professor in Family and Consumer Sciences, University of Georgia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2521RC296228
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Bone Health; Cognitive Health
Keywords: Bone; Cognition; Egg; Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole egg powder arm (Experimental): The whole egg powder arm will be part of our food product intervention. Food products created using whole egg powder will be provided and consumed 10x/week for 9 months. Each food item will contain the equivalent of one whole egg.
  Interventions: Other: Whole egg powder
- Whole milk powder arm (Active Comparator): The whole milk powder arm will be part of our food product intervention. Food products created using whole milk powder will be provided and consumed 10x/week for 9 months. These items will have the equivalent amount of protein as the whole egg group. They will be isocaloric in nature.
  Interventions: Other: Whole milk powder
- Gelatin arm (Placebo Comparator): The gelatin food products will be a part of our food product intervention. Food products created using gelatin will be provided and consumed 10x/week for 9 months. These items will be isocaloric in nature to the other treatment arms but will not contain additional protein.
  Interventions: Other: Gelatin food product

INTERVENTIONS:
Other: Whole egg powder — Participants will receive waffles, pancakes, brownies, ice cream and mac and cheese made with whole egg powder. The food projects were developed specifically for this study by the University of Georgia's Food Product Innovation and Commercialization Center and consumer tested by children within the study age range prior to intervention enrollment.
  Arms: Whole egg powder arm
Other: Whole milk powder — Participants will receive waffles, pancakes, brownies, ice cream and mac and cheese made with whole milk powder. The food projects were developed specifically for this study by the University of Georgia's Food Product Innovation and Commercialization Center and consumer tested by children within the study age range prior to intervention enrollment.
  Arms: Whole milk powder arm
Other: Gelatin food product — Participants will receive waffles, pancakes, brownies, ice cream and mac and cheese made with gelatin. The food projects were developed specifically for this study by the University of Georgia's Food Product Innovation and Commercialization Center and consumer tested by children within the study age range prior to intervention enrollment.
  Arms: Gelatin arm

SUMMARY:
This project is the first egg feeding randomized controlled trial (RCT) in children. The goal of this RCT is to determine if eating formulated whole egg products for 9 months improves bone health and cognitive function in children ages 9-13 years more than children consuming products made of milk powder or gelatin.

DETAILED DESCRIPTION:
This 9-month randomized controlled trial is an egg product intervention in otherwise healthy, 9-13 year-old children in the early stages of puberty (N=120). It will assess changes in bone material and geometric properties using dual energy x-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT). Cognitive function will be measured by the National Institute of Health's Toolbox. Participants will be randomized to one of 3 treatment (i.e., whole egg powder, whole milk powder, or gelatin) groups, and instructed to consume the food projects 10 times/week in substitute for other similar food products in their diet for 9-months. Five product choices per treatment group will be provided. The food products were developed specifically for this study by the University of Georgia's Food Product Innovation and Commercialization center and consumer tested. Additionally, these food products will be micro-tested prior to distribution to participants. We hypothesize that children consuming whole egg products will have enhanced bone outcomes and cognitive abilities in comparison to those consuming whole milk powder or gelatin.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy and well-nourished
* White, Black or Hispanic
* Males and females between the chronological ages of 9-13 years
* Sexual maturation rating, as measured by Tanner, at stages 2/3.
* Must be willing to provide a blood sample
* Not allergic to egg or egg products, milk or milk products, or gelatin

Exclusion Criteria:

* Achievement of menarche (females)
* Sexual maturation rating, as measured by Tanner, at stages 4/5
* Known bone disease or disease know to influence bone metabolism (e.g., cerebral palsy, intestinal malabsorption, juvenile rheumatoid arthritis)
* Known growth disorders
* The use of medications that may influence bone metabolism (e.g., corticosteroids, attention-deficit/hyperactivity disorder medications)
* Allergic to egg or egg products, milk or milk products, or gelatin

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

PRIMARY OUTCOMES:
Bone Outcomes | Assess changes in bone outcomes from baseline to 9 months
  Three-dimensional cortical and trabecular bone geometry measures will be assessed via pQCT at the tibia and radius. Outcome measures from the pQCT will include cortical and trabecular bone mineral density, cortical bone mineral area, total area, periosteal circumference, endosteal circumference, strength strain index, and bone strain index. DXA will be used to assess two-dimensional bone measurements at the lumbar spine, non-dominant hip, forearm, and total body.
Body Composition | Measure changes in body composition from baseline to 4.5 months and 9 months.
  Body composition measures (i.e., total body fat mass, fat-free soft tissue mass, and percent body fat) will be assessed by DXA.
Cognitive Health | Changes in cognitive function will be assessed from baseline to 4.5 and 9 months
  Cognitive health will be measured using the National Institute of Health's Toolbox. This toolbox for which validity evidence and national norms for children have been provided (Tulsky et al., 2013; Akshoomoff et al., 2014; Weintraub et al., 2013; Zelazo et al., 2013), will measure six cognitive domains: Executive Function, Episodic Memory, Working Memory, Attention, Language Ability, and Processing Speed.

SECONDARY OUTCOMES:
Serum Lipids | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in serum lipids
Insulin | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in serum insulin
Insulin like growth factor 1 | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in insulin like growth factor 1
Vascular endothelial growth factor | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in vascular endothelial growth factor
C-reactive protein | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in C-reactive protein
Monocyte chemoattractant protein 1 | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in monocyte chemoattractant protein 1
Interleukin 6 | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in interleukin 6
Tumor necrosis factor alpha | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in tumor necrosis factor alpha
Glucose | Serum samples will be collected at baseline, 4.5 months and 9 months
  Changes in glucose

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Lewis, PhD, Principal Investigator — University of Georgia; Nicole J Crenshaw, Study Director — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tulsky DS, Carlozzi NE, Chevalier N, Espy KA, Beaumont JL, Mungas D. V. NIH Toolbox Cognition Battery (CB): measuring working memory. Monogr Soc Res Child Dev. 2013 Aug;78(4):70-87. doi: 10.1111/mono.12035. PMID 23952203
- [Result] Akshoomoff N, Newman E, Thompson WK, McCabe C, Bloss CS, Chang L, Amaral DG, Casey BJ, Ernst TM, Frazier JA, Gruen JR, Kaufmann WE, Kenet T, Kennedy DN, Libiger O, Mostofsky S, Murray SS, Sowell ER, Schork N, Dale AM, Jernigan TL. The NIH Toolbox Cognition Battery: results from a large normative developmental sample (PING). Neuropsychology. 2014 Jan;28(1):1-10. doi: 10.1037/neu0000001. Epub 2013 Nov 11. PMID 24219608
- [Result] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Result] Zelazo PD, Anderson JE, Richler J, Wallner-Allen K, Beaumont JL, Weintraub S. II. NIH Toolbox Cognition Battery (CB): measuring executive function and attention. Monogr Soc Res Child Dev. 2013 Aug;78(4):16-33. doi: 10.1111/mono.12032. PMID 23952200
- [Derived] O'Connor PJ, Chen X, Coheley LM, Yu M, Laing EM, Oshri A, Marand A, Lance J, Kealey K, Lewis RD. The effects of 9 months of formulated whole-egg or milk powder food products as meal or snack replacements on executive function in preadolescents: A randomized, placebo-controlled trial. Am J Clin Nutr. 2022 Dec 19;116(6):1663-1671. doi: 10.1093/ajcn/nqac281. PMID 36173384